CLINICAL TRIAL: NCT02268786
Title: Prospective, Multi-center, Randomized Controlled Trial Comparing Pregnancy Outcomes Following Selection and Single Embryo Transfer (SET) Based on Preimplantation Genetic Screening (PGS) by Next Generation Sequencing (NGS) Versus Standard Morphological Assessment
Brief Title: Single Embryo TrAnsfeR of Euploid Embryo
Acronym: STAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Illumina, Inc. (Industry)
Collaborators: Reprogenetics (Industry); Genesis Genetics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: RGH-001
Record Dates: First submitted 2014-10-15; First posted 2014-10-20 (Estimated); Results first posted 2020-05-04 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Infertility; Aneuploidy
Keywords: Preimplantation Genetic Screening; Blastocyst; Vitrification; In vitro fertilization; non-invasive prenatal testing; next generation sequencing
MeSH Terms: conditions — Infertility; Aneuploidy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Intent to transfer single euploid embryo based on NGS testing (VeriSeq™ PGS) of biopsied blastocysts
  Interventions: Other: Preimplantation Genetic Screening by NGS
- Group B (No Intervention): Intent to transfer single embryo based on morphological assessment according to the Gardner scoring system (no PGS)

INTERVENTIONS:
Other: Preimplantation Genetic Screening by NGS — The VeriSeq PGS takes advantage of next-generation sequencing (NGS) technology to provide comprehensive, accurate screening of all 24 chromosomes for selection of euploid embryos.
  Other Names: Veriseq PGS
  Arms: Group A

SUMMARY:
The purpose of the current study is to evaluate the effect of preimplantation genetic screening (PGS) by next generation sequencing (NGS) compared to standard morphological assessment of embryos on pregnancy rates through a randomized controlled trial (RCT). All embryos will be vitrified and a single embryo transfer (SET) will be performed with either screened or unscreened embryos depending on randomization.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing IVF
* At least 2 blastocysts suitable for biopsy on day 5 or 6 of embryo development

Exclusion Criteria:

* History of more than two prior implantation failure following IVF
* History of more than one miscarriage of viable pregnancy
* One or both partners known to be carrier(s) of a chromosomal abnormality
* Known genetic carrier couple and/or one or both partners carrier of a known autosomal dominant disorder
* Any other non-study related preimplantation genetic testing
* Use of donor oocytes
* Use of gestational carrier (surrogate or donor egg recipient).
* Severe oligospermia (<1,000,000 sperm/ml); Surgical Sperm Retrieval for reasons other than post-vasectomy and CAVD
* Low ovarian reserve with (FSH) >10 IU/L on day 2-4 of a prior menstrual cycle and/or (AMH) <7 pmol/L (or <1 ng/ml)
* Gender selection cycles
* Concurrent participation in another clinical trial

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 661 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (38):
- United States (28):
  - Fertility Treatment Center, Tempe, Arizona
  - HRC Fertility, Encino, California
  - Acacio Fertility Clinic, Laguna Niguel, California
  - HRC Fertility Pasadena, Pasadena, California
  - Fertility Specialists Medical Group, San Diego, California
  - Reproductive Science Center of San Francisco Bay Area, San Ramon, California
  - Colorado Center for Reproductive Medicine (CCRM), Lonetree, Colorado
  - Reproductive Associates of Delaware, Newark, Delaware
  - CRM Orlando, Orlando, Florida
  - Georgia Reproductive Specialists, Atlanta, Georgia
  - Fertility Institute of Hawaii, Honolulu, Hawaii
  - Fertility Center of Illinois, Highland Park, Highland Park, Illinois
  - The Advanced IVF Institute, Naperville, Illinois
  - IVF New England, Lexington, Massachusetts
  - IVF Michigan, Bloomfield Hills, Michigan
  - Genesis Genetics (USA) - Genetics Laboratory, Plymouth, Michigan
  - Reproductive Science Center of New Jersey, Eatontown, New Jersey
  - Reprogenetics (USA) - Genetics Laboratory, Livingston, New Jersey
  - IRMS at St. Barnabas, Livingston, New Jersey
  - Main Line Fertility, Bryn Mawr, Pennsylvania
  - Texas Fertility Center, Austin, Texas
  - Dallas Fertility Center, Dallas, Texas
  - Dallas IVF, Frisco, Texas
  - Houston Fertility Institute, Houston, Texas
  - CORM Houston, Webster, Texas
  - Utah Fertility Center, Pleasant Grove, Utah
  - Reproductive Care Center, Sandy City, Utah
  - Seattle Reproductive Medicine, Seattle, Washington
- Melbourne IVF, Melbourne, Victoria, Australia
- Canada (3):
  - Olive Fertility Centre, Vancouver, British Columbia
  - Reproductive Care Center, Mississauga, Ontario
  - TRIO Fertility Treatment Practice, Toronto, Ontario
- United Kingdom (6):
  - Boston Place Clinic, London, Greater London
  - Care Fertility Group London, London, Greater London
  - Care Fertility Group Manchester, Manchester, Greater Manchester
  - Oxford Fertility Unit, Oxford, Oxfordshire
  - Genesis Genetics (UK) - Genetics Laboratory, London
  - Reprogenetics (UK) - Genetics Laboratory, Oxford

REFERENCES:
- [Result] Handyside AH. 24-chromosome copy number analysis: a comparison of available technologies. Fertil Steril. 2013 Sep;100(3):595-602. doi: 10.1016/j.fertnstert.2013.07.1965. PMID 23993662
- [Result] Schoolcraft WB, Katz-Jaffe MG. Comprehensive chromosome screening of trophectoderm with vitrification facilitates elective single-embryo transfer for infertile women with advanced maternal age. Fertil Steril. 2013 Sep;100(3):615-9. doi: 10.1016/j.fertnstert.2013.07.1972. PMID 23993664
- [Result] Yang Z, Liu J, Collins GS, Salem SA, Liu X, Lyle SS, Peck AC, Sills ES, Salem RD. Selection of single blastocysts for fresh transfer via standard morphology assessment alone and with array CGH for good prognosis IVF patients: results from a randomized pilot study. Mol Cytogenet. 2012 May 2;5(1):24. doi: 10.1186/1755-8166-5-24. PMID 22551456
- [Result] Fiorentino F, Biricik A, Bono S, Spizzichino L, Cotroneo E, Cottone G, Kokocinski F, Michel CE. Development and validation of a next-generation sequencing-based protocol for 24-chromosome aneuploidy screening of embryos. Fertil Steril. 2014 May;101(5):1375-82. doi: 10.1016/j.fertnstert.2014.01.051. Epub 2014 Mar 6. PMID 24613537
- [Result] Bianchi DW, Parker RL, Wentworth J, Madankumar R, Saffer C, Das AF, Craig JA, Chudova DI, Devers PL, Jones KW, Oliver K, Rava RP, Sehnert AJ; CARE Study Group. DNA sequencing versus standard prenatal aneuploidy screening. N Engl J Med. 2014 Feb 27;370(9):799-808. doi: 10.1056/NEJMoa1311037. PMID 24571752
- [Result] Munne S, Kaplan B, Frattarelli JL, Child T, Nakhuda G, Shamma FN, Silverberg K, Kalista T, Handyside AH, Katz-Jaffe M, Wells D, Gordon T, Stock-Myer S, Willman S; STAR Study Group. Preimplantation genetic testing for aneuploidy versus morphology as selection criteria for single frozen-thawed embryo transfer in good-prognosis patients: a multicenter randomized clinical trial. Fertil Steril. 2019 Dec;112(6):1071-1079.e7. doi: 10.1016/j.fertnstert.2019.07.1346. Epub 2019 Sep 21. PMID 31551155
- [Derived] Cornelisse S, Zagers M, Kostova E, Fleischer K, van Wely M, Mastenbroek S. Preimplantation genetic testing for aneuploidies (abnormal number of chromosomes) in in vitro fertilisation. Cochrane Database Syst Rev. 2020 Sep 8;9(9):CD005291. doi: 10.1002/14651858.CD005291.pub3. PMID 32898291

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Genetic Screening by NGS: Group A: Genetic Screening by NGS (PGT-A)
- Group B: Morphology Only: Group B: Morphology Only (Control)
Period: Overall Study
Arm/Group | Group A: Genetic Screening by NGS | Group B: Morphology Only
Started | 330 | 331
Completed | 274 | 313
Not Completed | 56 | 18
Not completed — No Euploid Embryos available | 42 | 0
Not completed — Withdrawal by Subject | 7 | 14
Not completed — Thaw Failure | 6 | 4
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Genetic Screening by NGS | Group B: Morphology Only | Total
Number analyzed (Participants) | 330 | 331 | 661
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 330 | 331 | 661
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.7 (3.59) | 33.8 (3.58) | 33.7 (3.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 330 | 331 | 661
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 42 | 32 | 74
  United States | 244 | 244 | 488
  United Kingdom | 34 | 43 | 77
  Australia | 10 | 12 | 22

OUTCOME MEASURES:

1. Primary Outcome: Ongoing Pregnancy
Description: Number of Participants with Ongoing Pregnancy at 20 Weeks Gestation
Time Frame: Gestational Age of 20 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Genetic Screening by NGS | Group B: Morphology Only
Number analyzed (Participants) | 274 | 313
Participants | 137 | 143

ADVERSE EVENTS:
Arm/Group | Group A: Genetic Screening by NGS | Group B: Morphology Only
Serious Adverse Events (participants affected / at risk) | 0/330 | 0/331
Other Adverse Events (participants affected / at risk) | 0/330 | 0/331

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days